CLINICAL TRIAL: NCT03308110
Title: A PHASE 1, SINGLE DOSE, OPEN LABEL, RANDOMIZED, 5-PERIOD CROSSOVER STUDY TO EVALUATE THE RELATIVE BIOAVAILABILITY AND FOOD EFFECT ON NEW MODIFIED RELEASE TABLET OF PF-06650833 IN HEALTHY SUBJECTS
Brief Title: Bioavailability and Food Effect Study of Two Formulations of PF-06650833
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B7921011; 2017-002052-88 (EudraCT Number)
Record Dates: First submitted 2017-09-05; First posted 2017-10-12 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — 1-(((2S,3S,4S)-3-ethyl-4-fluoro-5-oxopyrrolidin-2-yl)methoxy)-7-methoxyisoquinoline-6-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relative Bioavailability Cohort (Other): Relative Bioavailability cohort
  Interventions: Drug: PF-06650833

INTERVENTIONS:
Drug: PF-06650833 — Two formulations of PF-006650833

SUMMARY:
Bioavailability and food effect of 2 formulations of PF-06650833 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of nonchild bearing potential and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Subjects with any of the following characteristics/conditions will not be included in the study:

Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

Any condition possibly affecting drug absorption (eg, gastrectomy).

* A positive urine drug test.
* History of regular alcohol consumption within 6 months before screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product (whichever is longer).
* Screening supine BP greater than equal to 140 mm Hg (systolic) or more than equal to 90 mm Hg (diastolic), following at least 5 minutes of supine rest.
* Pregnant female subjects; breastfeeding female subjects; female subjects of childbearing potential;
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product.
* History of tuberculosis or active or latent or inadequately treated infection, positive QuantiFERON-TB Gold test.

History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb).

-Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-96 hours
AUClast | 0-96 hours

SECONDARY OUTCOMES:
Cmax under high fat meal fed conditions | 0-96 hours
Pharmacokinetic parameters of PF-06650833 from plasma concentration (if data permits) | 0-96 hours
AUClast under high fat meal fed conditions | 0-96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7921011&StudyName=A+Phase+1%2C+Single+Dose%2C+Open+Label%2C+Randomized%2C+5-period+Crossover+Study+To+Evaluate+The+Relative+Bioavailability+And+Food+Effect+On+New+Modified+Release+Tablet+Of+Pf-06650833+In+Healthy+Subjects